CLINICAL TRIAL: NCT05554159
Title: A Virtually Delivered Exercise Intervention To Mitigate Cognitive Deficits From Radiotherapy In AYAs With Brain Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0152; NCI-2022-08000 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Brain Tumor; Brain Cancer
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Actigraph (Experimental): A device worn on the waist that measures physical activity (such as the number of steps participants walk each day, how long participants spend standing, and how long partticipants spend laying down). Participants should wear the ActiGraph at least 10 hours a day for 7 days.
  Interventions: Behavioral: Standard Fitbit Program; Behavioral: Virtual Exercise Program

INTERVENTIONS:
Behavioral: Standard Fitbit Program — Participants will be given a Fitbit to wear during their participation in this program. Participants will need to wear the Fitbit at least 5 days per week and for at least 10 hours a day. Participants will take part in video calls (through the video conferencing platform Zoom) 1 time a week.
Behavioral: Virtual Exercise Program — Participants will be given a Fitbit to wear during their participation in this program. Participants will need to wear the Fitbit at least 5 days per week and for at least 10 hours a day. Participants will take part in video calls (through the video conferencing platform Zoom) 1 time a week.

SUMMARY:
To test a new investigational virtual exercise program for adolescents and young adults (AYAs) with brain tumors who plan to receive cranial radiotherapy

DETAILED DESCRIPTION:
Primary Objective:

Determine the feasibility and acceptability of a virtually supervised exercise intervention compared to control in AYAs with brain tumors undergoing cranial radiotherapy (CRT).

Secondary Objective:

Assess the effect of supervised exercise intervention on the neuroanatomic structure and cognitive function changes in AYAs with brain tumors undergoing CRT.

Exploratory Objective:

Assess the effect of supervised exercise intervention on other brain structure (white matter integrity), cognitive functions (attention, visual learning, psychomotor function, executive function, verbal learning, working memory and clinician-reported neurological exam outcomes), patient-reported health-related quality of life, objectively measured and patient-reported physical activity level, patient-reported dietary recall, objectively measured physical function assessments, and exercise progression (exercise volume). Assess the agreement between physical function tests performed twice virtually.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15-39 years old
2. Self-reported diagnosis of a primary benign or malignant brain tumor or confirmed diagnosis of primary benign or malignant brain tumor radiographically or pathologically when available (relapse or newly diagnosed)
3. Plans to receive CRT at MDACC or, if the participant has already started CRT, the participant is eligible if they are within 3 weeks of the start of CRT
4. Received appropriate physician clearance
5. Able to move arms and legs, and ambulate safely
6. Participant is insufficiently active (reports less than 150 minutes of planned moderate-vigorous intensity activity per week in the prior week)
7. Participants and/or guardians are willing and able to provide informed consent
8. Has a smartphone with available space to download additional apps
9. Does not have sensorimotor strip impairment as indicated by the clinical team
10. Has internet access
11. Can receive physical therapy because this is part of the standard of care
12. Participants and/or guardians are willing and able to provide informed consent for protocol PA18-0130 (Pediatric Energy Balance Data Repository Study), companion protocol for the Fitbit application/assessment.

Exclusion Criteria:

1. Non-English speaking
2. Screen failure for exercise safety based on Physical Activity Readiness Questionnaire (PAR-Q).12
3. Underlying unstable cardiac or pulmonary disease or symptomatic cardiac disease
4. Recent fracture or acute musculoskeletal injury that precludes ability to participate in supervised exercise training sessions
5. Cognitive and/or major sensory deficits that would impede the completion of research activities and assessments as deemed by the clinical team.
6. Self-reported diagnosis of a metastatic brain tumor or confirmed diagnosis of a metastatic brain tumor radiographically or pathologically when available
7. Self-report of pregnancy
8. Currently enrolled in another physical activity or exercise intervention
9. Prisoners
10. Self-reported pregnancy status

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
MD Anderson Symptom Inventory - Brain Tumor (MDASI - BT) | Through study completion an average of 1 year.
  Scale Score ranges from 0-10
  0-Symptom has not been present 10-The symptom was as bad as you can imagine it could be

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Schadler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-04-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT05554159/ICF_000.pdf